CLINICAL TRIAL: NCT05569902
Title: Remember NIBS? tACS Improves Memory Performance in Elders With Subjective Memory Complaints
Brief Title: tACS Improves Memory in Elders With Subjective Memory Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, reza kazemi, Assistant professor, University of Tehran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tACS
Record Dates: First submitted 2022-09-24; First posted 2022-10-06 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Memory Deficits; tACS
Keywords: Episodic memory; medial Prefrontal Cortex; tACS; SMC
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tACS (Experimental): Participants in this group received 20 minutes of active 6 Hz stimulation over the medial prefrontal cortex.
  Interventions: Device: active tACS
- Sham tACS (Sham Comparator): Participants in this group received 20 minutes of sham stimulation over the medial prefrontal cortex.
  Interventions: Device: sham tACS

INTERVENTIONS:
Device: active tACS — transcranial alternating current stimulation is a non-invasive method of entraining specific frequency bands in the brain by applying weak intensities of electric current in a desired shape and phase to the desired brain regions.
  Arms: Active tACS
Device: sham tACS — transcranial alternating current stimulation is a non-invasive method of entraining specific frequency bands in the brain by applying weak intensities of electric current in a desired shape and phase to the desired brain regions.
  Arms: Sham tACS

SUMMARY:
Subjective memory complaints (SMC), the main cognitive component of which is event memory, is a predictor of Alzheimer's disease in elderly people. The purpose of this study was to investigate the effect of transcranial alternating current stimulation (tACS) with theta frequency (6 Hz) on the medial prefrontal cortex in the improvement of episodic memory in individuals with SMC in a double blind, randomized, and sham-controlled parallel study. Sixteen participants with SMC received either active or sham theta tACS on the medial prefrontal cortex (mPFC). EEG was recorded and Rey Auditory Verbal Learning Test (RAVLT) was administered. The aim of the current study was to see if theta tACS over the mPFC can improve event memory in individuals with SMC and thus can be considered a potential therapeutic intervention for this population or not.

ELIGIBILITY:
Inclusion Criteria:

* Being 50 or older,
* Mini Mental State Examination (MMSE) grade from 27 to 30
* Total score of 58 or more on the Everyday Memory Questionnaire (EMQ)
* no indications of depression and anxiety measured by Geriatric Depression Scale (GDS) and State-Trait Anxiety Inventory (STAI)
* No sign of dementia based on Diagnostic and statistical manual of mental disorder, 5th edition (DSM-V) criteria

Exclusion Criteria:

* History of a major psychological or neurological condition
* History of head trauma leading to unconsciousness,
* Presence of metal in the head
* History of seizures
* Serious cardiovascular disease
* Use of medications with an impact on cognitive functions
* Recent use of alcohol or substance abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in performance | 25 minutes i.e., before versus after the stimulation
  Rey auditory-verbal learning test (RAVLT)

SECONDARY OUTCOMES:
Change in EEG power in theta frequency band | 30 minutes, i.e., before versus after stimulation
  Spectral analysis measuring power in different frequency bands
Change in phase synchronization connectivity in theta frequency band | 30 minutes, i.e., before versus after stimulation
  Phase relations between neural signals realized by means of phase-locking values (PLV)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Rostami, M.D., Study Director — University of Tehran; Sahereh Varastegan, MSc, Principal Investigator — University of Tehran
Locations (1):
- National Brain Mapping Lab, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No